CLINICAL TRIAL: NCT00693537
Title: Long- But Not Short-term Exercise Training Improves Coronary Endothelial Dysfunction in Diabetes Mellitus Type 2 and Coronary Artery Disease
Brief Title: Exercise Training Improves Coronary Endothelial Dysfunction in Diabetes Mellitus Type 2 and Coronary Artery Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Prof. Josef Niebauer M.D., Ph.D., MBA, Director of Institute, Paracelsus Medical University
Allocation: Randomized
Other Study IDs: UISM-2-2008
Record Dates: First submitted 2008-06-04; First posted 2008-06-09 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2008-06

CONDITIONS: Type 2 Diabetes Mellitus; Coronary Artery Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease | interventions — Exercise

ARMS (2):
- A (Experimental): 4 weeks in-hospital exercise training (6x15 min bicycle/day, 5 days/week) followed by a 5 months ambulatory exercise program (30 min ergometer/day, 5 days/week, plus 1h group exercise/week)
  Interventions: Behavioral: Exercise training
- B (No Intervention): Control

INTERVENTIONS:
Behavioral: Exercise training — 4 weeks in-hospital exercise training (6x15 min bicycle/day, 5 days/week) followed by a 5 months ambulatory exercise program (30 min ergometer/day, 5 days/week, plus 1h group exercise/week)
  Arms: A

SUMMARY:
Patients with type 2 diabetes mellitus suffer from accelerated coronary artery disease. We will assess the effects of exercise training on coronary endothelial function, vascular structure, and inflammation both in serum and skeletal muscle biopsies, as well as expression of diabetes candidate genes.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* preserved left ventricular function (left ventricular ejection fraction ≥ 50%)
* a physical work capacity ≥ 50 W
* at least one significant coronary stenosis > 50%, whereas either the left anterior descending (LAD) or circumflex artery (RCX) has to be free from disease or stenoses ≤ 25% for the assessment of intracoronary flow measurements

Exclusion Criteria:

* diseases further affecting endothelial function
* untreated hypertension (systolic blood pressure > 160 mm Hg or a diastolic blood pressure of > 90 mm Hg)
* cigarette smoking during the previous six months
* LDL-cholesterol > 4.3 mmol/l
* ventricular tachyarrhythmias
* chronic obstructive pulmonary disease
* severe renal or hepatic dysfunction
* valvular heart disease
* myocardial infarction within the previous 4 weeks

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University Institute of Sports Medicine, Prevention and Rehabilitation, Salzburg, Austria